CLINICAL TRIAL: NCT02360930
Title: The Pharmacokinetics and Pharmacodynamics of Vincristine in the Adolescent and Young Adult Population Compared to Younger Children
Brief Title: Vincristine PK and PD in the AYA Population Compared to Younger Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Leidy Isenalumhe, Hematology-Oncology Fellow, Children's Hospital Los Angeles
Other Study IDs: CHLA CCI-14-00092
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Leukemia, Acute Lymphoblastic; Leukemia
Keywords: Acute Lymphoblastic Leukemia; Pharmacokinetics; Vincristine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tanner Stage </=2: Patients will be stratified by phase of treatment, and they will be classified into Tanner stage ≤ 2 or ≥ 4, based on physical examination. We plan to have 15 patients in Tanner staging ≤ 2 and 15 patients in Tanner staging ≥ 4.
- Tanner Stage >/= 4: Patients will be stratified by phase of treatment, and they will be classified into Tanner stage ≤ 2 or ≥ 4, based on physical examination. We plan to have 15 patients in Tanner staging ≤ 2 and 15 patients in Tanner staging ≥ 4.

SUMMARY:
The trial is to determine if a difference exists in the way that adolescents and young adults metabolize the chemotherapy agent vincristine compared to younger children.

DETAILED DESCRIPTION:
The purpose of the study is to refine the PK model for planning a future definitive study. This is a pilot study to obtain preliminary data on the pharmacokinetics of VCR and the way it differs in the AYA population compared to the younger children as defined by Tanner staging. Additionally, we want to determine if Calpain levels correlate with vincristine and its PK and to determine if it can be used as biomarker for VRNT.

Specific Aim 1: Develop a non-parametric population model of vincristine and M1 PK in children and adolescents.

Hypothesis: The PK of vincristine and its metabolite M1 will differ between young children and AYA as defined by Tanner stage

Specific Aim 2: Measure repeated serum calpain with initiation of vincristine and again after four weeks of therapy.

Hypothesis: Compared to baseline, serum calpain will increase after administration of vincristine.

For the first time, patients will be classified based on their physiologic maturity-rather than age-to determine whether having a more adult phenotype is associated with prolonged vincristine exposure. This will increase our likelihood of detecting a developmentally-driven difference in vincristine metabolism and, if successful, provide evidence that Tanner staging is a more reliable method for classifying adolescents for purposes of chemotherapy dosing. Further, we will not only characterize vincristine PK differences between the two groups, but will for the first time examine differences in the PK of M1.We are analyzing calpain levels as a separate entity from Tanner staging. We are trying to establish if there is an association between calpain and vincristine administration, as well as vincristine induced peripheral neuropathy. However, in evaluating the association between vincristine dose, PK and calpain levels, we will be adjusting for age and Tanner stage in the analysis.

To account for enzyme polymorphism in the metabolism of vincristine, we will analyze each patient for CYP3A5 genotype, which has been associated with increase in clearance of vincristine and less peripheral neuropathy and decrease severity of vincristine induced peripheral neuropathy. Additionally, we will determine the vincristine's PK which will allow us to probe the impact of polymorphism with regards to VCR disposition.

For all of the following aims, we will enroll a total of 30 patients with a unified diagnosis of acute lymphoblastic leukemia (ALL),6 months to 21 in Induction phase or in Maintenance phase of therapy. Patients will be stratified by phase of treatment, and they will be classified into Tanner stage ≤ 2 or ≥ 4, based on physical examination. We plan to have 15 patients in Tanner staging ≤ 2 and 15 patients in Tanner staging ≥ 45. Each patient will receive vincristine weekly x 4 (Induction) or monthly (Maintenance), at a standard dose specified by the treatment protocol. Since PK measurements will be obtained around a single VCR dose; it is appropriate to include patients with ALL from two phases of treatment. The study will be conducted at a single institution, Children's Hospital Los Angeles (CHLA). From the newly diagnosed patients in Induction phase, we will collect optimally timed blood samples prior to and 10 minutes, 30 minutes, 1 hour, 12 hours and 24 hours following the first dose of vincristine. We will also measure serum calpain, a candidate biomarker for nerve injury, before and after the first dose of vincristine, and again after the 4th weekly dose. For the ALL patients in the Maintenance phase, we will collect optimally timed blood samples prior to and 10 minutes, 30 minutes, 1 hours and 24 hours following the dose of vincristine. In ALL patients in Maintenance, a 12 hour blood sample will not be feasible since these patients are treated in the outpatient setting. We will also measure serum calpain levels prior to vincristine dose, 24 hours after and 4 weeks after the measured vincristine level. The study period for ALL patients in Maintenance phase will be completed 4 weeks after initial measured VCR PK level.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 1-24 years of age with Acute Lymphoblastic Leukemia
* Patient diagnosed with Acute Lymphoblastic Leukemia (ALL) in Induction phase of therapy
* Patient diagnosed with Acute Lymphoblastic Leukemia (ALL) in first remission in Maintenance phase of therapy Treatment plan for induction therapy includes vincristine given at weekly intervals.
* Treatment plan for Maintenance therapy includes vincristine given at monthly intervals.

Exclusion Criteria:

* Patients without a central line in induction phase of therapy

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 30 patients with ALL. Our study will enroll patients ages 1-24 years with ALL at start of Induction or in Maintenance therapy. Patients will be classified into Tanner stage ≤ 2 or ≥ 4. We plan to have 15 patients in Tanner staging ≤ 2 and 15 patients in Tanner staging ≥ 4. Each patient will receive vincristine weekly x 4 (Induction) or monthly (Maintenance), at a standard dose specified by the treatment protocol.
  The study will be conducted at Children's Hospital Los Angeles.
  Tanner staging will take place after the patient is consented to the study using standard Tanner stage diagrams.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Vincristine (concentration of vincristine) | 4 weeks
  We will evaluate the concentration of vincristine in relations to the production of primary metabolite M1 over time. Vincristine is primary metabolized using CYP3A family of enzymes is responsible.

SECONDARY OUTCOMES:
Calpain level | 4 weeks
  Serum calpain enzyme activity will be measured at three time points: 1) just prior to the first dose of vincristine to establish baseline levels; 2) 24 hours after the first dose of vincristine to measure acute effects of vincristine on enzyme activity; 3) after the 4th weekly vincristine (Induction) or after 4 weeks since last VCR dose (Maintenance) to assess chronic effects
Cytochrome P450 3A5 genotype | One time
  One whole blood sample will be collected for DNA extraction and genotyping from each subject enrolled in this study.
Development of Vincristine Induced Neuropathy | 4 weeks
  To screen for development of VRNT, we will employ two validated measures, the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE 4.0)24 and the Pediatric-Modified Total Neuropathy Score.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Damerla, Study Director — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States